CLINICAL TRIAL: NCT02517346
Title: Efficacy of Telemonitoring on CPAP Treatment Compliance in Obstructive Sleep Apnea (OSA) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: ResMed (Industry); Asociacio Lleidatana de Respiratori (Unknown)
Responsible Party: Principal Investigator, Ferran Barbe, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SEPAR2015
Record Dates: First submitted 2015-07-30; First posted 2015-08-07 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2015-08

CONDITIONS: Sleep Apnea Syndrome
Keywords: CPAP compliance; Telemonitoring; Standard management; Cost effectiveness
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard follow up-Sleep Unit (Active Comparator): Patients diagnosed as OSA, treated with CPAP and followed up in sleep unit
  Interventions: Other: Standard follow-up
- Telemonitoring (Experimental): Patients diagnosed as OSA and treated with CPAP in sleep unit, followed up by telemonitoring system
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Standard follow-up — Standard management according to Spanish Respiratory Society guidelines in Sleep Unit.
  Arms: Standard follow up-Sleep Unit
Other: Telemonitoring — Follow up by telemonitoring system during 3 months
  Arms: Telemonitoring

SUMMARY:
The purpose of this study is to compare the effectiveness of telemonitoring versus standard follow-up on CPAP treatment compliance in Obstructive Sleep Apnea Syndrome (OSAS).

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is defined by the presence of repetitive episodes of upper airways collapse during sleep, leading to nocturnal hypoxemia, sleep fragmentation and daytime sleepiness. When untreated, OSA is a risk factor for arterial hypertension , cardiovascular and cerebrovascular diseases, road accidents and a worse quality of life. The application of a continuous positive airways pressure (CPAP) represents the first line therapy in patients with moderate to severe OSA. CPAP treatment improves daytime sleepiness and oxygen saturation , reduces cardiovascular risk, ameliorates neurobehavioral performance, improves quality of life and reduces road accidents. Despite its demonstrated efficacy, CPAP effectiveness is significantly limited by poor adherence. A closer follow up could improve CPAP adherence but it would take up more work and additional costs for sleep units.

So on that account, the investigators propose a study to demonstrate that automatic home treatment monitoring of patients with OSA is a cost-effectiveness alternative approach to patient's management. Moreover, the investigators believe that telemonitoring could improve CPAP compliance and patient's satisfaction and reduce follow-up costs.

Methods:

Prospective and randomized study during three months. Patients diagnosed as OSA in St. Maria's Hospital (Sleep Unit) and requiring CPAP treatment, will be randomized into two groups differing in CPAP compliance monitoring and management .

Group 1 Standard care Patients will be fitted with a mask and given a CPAP and instructed on how to use the device. Patients will follow the standard treatment management. All patients will be visited at 1 month at sleep unit. Patients will be checked about progress and adherence to therapy and any problems with their machine. Information will be downloaded from their machines (CPAP adherence, applied CPAP pressure, mask leak, and residual respiratory events…).

Group 2 Telemonitoring Patients will be fitted with a mask and given a CPAP. Each CPAP device will be provided with a modem sending daily compliance information (CPAP adherence, CPAP pressure, mask leak, and residual respiratory events) to a web database.

Patients of both 2 groups will be finally visited at 3 months at sleep unit.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women over 18 years old
* Diagnosed as OSA and requiring CPAP treatment
* Written informed consent form signed.

Exclusion Criteria:

* Patients with impaired lung function (overlap syndrome, obesity hypoventilation syndrome, and restrictive disorders)
* Severe heart failure
* Severe chronic pathology associated
* Psychiatric disorder
* Periodic leg movements
* Pregnancy
* Other dyssomnias or parasomnias
* Patients already treated with CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
CPAP adherence at 3 months | 3 months
  Number of hours of use per day of CPAP according to the internal clock of the CPAP device

SECONDARY OUTCOMES:
Patients' satisfaction at 3 months | 3 months
  Patients will be asked to grade their satisfaction with the follow up care provided by telemonitoring /sleep unit using a questionnaire and a visual analogue scale.
Cost effectiveness at 3 months | 3 months
  Costs in each group (CPAP carrying charge, number of visits and calls, number of hospital admissions) will be compared.
Change from baseline in quality of life at 3 months | 3 months
  EuroQOL health questionnaire and visual analogue scale will be used.
Fast detection of the non-adherent patient with telemonitoring | 3 months
  We assume that telemonitoring could quickly detect non- adherent patients.
Change in blood pressure at 3 months | 3 months
Change in body mass index at 3 months | 3 months
Abandons at 3 months | 3 months
  Number of patients lost at follow up at 3 months of CPAP therapy.
Adverse events at 3 months | 3 months
Change from baseline in snoring at 3 months | 3 months
  Patients will be asked about the persistence of snoring
Change from baseline in witnessed apneas at 3 months | 3 months
  Patients will be asked about the persistence of witnessed apneas
Change from baseline in nocturia at 3 months | 3 months
  Patients will be asked about the presence of nocturia.
Change from baseline in daytime sleepiness at 3 months | 3 months
  Epworth sleepiness scale will be used.
Changes in nocturnal gasping at 3 months | 3 months
  Patients will be asked about the persistence of nocturnal gasping
Changes in sleep fragmentation at 3 months | 3 months
  Patients will be asked about the persistence of sleep fragmentation/maintenance insomnia
Presence of symptoms of restlees leg syndrome at 3 months | 3 months
  Patients will be asked about the presence of symptoms of restless leg syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbe, MD, Principal Investigator — Hospital Arnau de Vilanova. IRB Lleida. CIBERes
Locations (1):
- Hospital Arnau de Vilanova-Santa María, Lleida, Lleida, Spain

REFERENCES:
- [Derived] Turino C, de Batlle J, Woehrle H, Mayoral A, Castro-Grattoni AL, Gomez S, Dalmases M, Sanchez-de-la-Torre M, Barbe F. Management of continuous positive airway pressure treatment compliance using telemonitoring in obstructive sleep apnoea. Eur Respir J. 2017 Feb 8;49(2):1601128. doi: 10.1183/13993003.01128-2016. Print 2017 Feb. PMID 28179438